CLINICAL TRIAL: NCT07281261
Title: Study of Transcutaneous Auricular Neurostimulation as a Treatment for Substance Use Disorder
Brief Title: tAN for Substance Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: The Menninger Clinic (Unknown); Baylor College of Medicine (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBM-AUD-01; H-56001 (Other: Baylor College of Medicine); R41AA032157 (NIH)
Record Dates: First submitted 2025-12-04; First posted 2025-12-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse; Substance Use Disorders; Substance Use Disorders Alcohol Use Withdrawal State
Keywords: Alcohol; Alcohol Use Disorder; Substance Use Disorder; Transcutaneous Auricular Neurostimulation; tAN; Neurostimulation; Vagus Nerve Stimulation; Auricular Neurostimulation; Transcutaneous
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, single-blind, sham-controlled trial. Participants will be randomized in a 1:1 ratio to one of two treatment groups: (1) Active tAN and (2) Sham tAN
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tAN (Experimental): Participants will have the device applied on-site (at the Menninger Clinic) and will be required to wear the device for a minimum of 4 hours of stimulation per day. Study assessments will be collected at the time of, prior to, and at the conclusion of each tAN treatment session. Active tAN stimulation will be administered in addition to the participant's standard of care treatment.
  Interventions: Device: Sparrow Ascent
- Sham tAN (Sham Comparator): Participants will have the device applied on-site (at the Menninger Clinic) and will be required to wear the device for a minimum of 4 hours of stimulation per day. Study assessments will be collected at the time of, prior to, and at the conclusion of each sham tAN treatment session. Sham tAN stimulation will be administered in addition to the participant's standard of care treatment.
  Interventions: Device: Sparrow Ascent (Sham)

INTERVENTIONS:
Device: Sparrow Ascent — The Sparrow Ascent is an FDA-cleared (K230796) wearable, battery-operated, neurostimulation system designed to transcutaneously stimulate nerves on and around the auricle. The system is comprised of a Patient Controller, cable, and 24-hour disposable earpiece.
  Other Names: Transcutaneous Auricular Neurostimulation
  Arms: Active tAN
Device: Sparrow Ascent (Sham) — Participants will have the earpiece applied and the cable connected to the Patient Controller, but tAN stimulation will not be turned on. The sham device has an identical appearance to the active device.
  Other Names: Transcutaneous Auricular Neurostimulation (Sham)
  Arms: Sham tAN

SUMMARY:
The study will involve a 5-day tAN treatment to attenuate alcohol withdrawal syndrome (AWS) and alter resting state functional connectivity (RSFC) between OFC and striatum in patients with alcohol use disorder (AUD). Enrolled participants will wear the tAN device on-site (at The Menninger Clinic) for the 5-day detox treatment period. Participants with AUD will be single-blinded randomized into 2 groups - a treatment group (active tAN) and a placebo group (sham tAN). Each group will consist of five separate time points - admission, screening, baseline, tAN treatment, and post tAN treatment. Clinical measures collected before, during, and after treatment will include alcohol withdrawal severity, craving, benzodiazepine usage, and assessments of depression and suicidal behaviors. Participants will undergo MRI scans before and after the treatment period to assess changes in brain connectivity and their relationship to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (evenly recruited) aged 18-64 years old
2. Meeting DSM-5 criteria of moderate or above AUD at screening using the structured clinical interview for DSM-5 (SCID-5)
3. Demonstration of at least moderate risk of alcohol use at screening using the WHO-ASSIST
4. Demonstration of high risk for moderate to severe alcohol withdrawal syndrome (Prediction of Alcohol Withdrawal Severity Scale [PAWSS] > 4 at admission)
5. Demonstration of severe withdrawal symptoms (Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised [CIWA-Ar] > 15 at screening)
6. Positive urine test for alcohol at screening
7. Be able to provide written informed consent
8. Female subjects must be non-nursing and not pregnant
9. Meet the MRI safety screening form provided by the Center for Advanced MR Imaging (CAMRI) at BCM.

Exclusion Criteria:

1. In the opinion of the clinician and the research team at admission, be expected to fail to complete the study protocol due to probably relocation from The Menninger Clinic area or not tolerable to receive tAN
2. Current use of tobacco
3. Is pregnant or nursing
4. Contraindications to MRI (pacemaker, cochlear implants, metal in eyes, other metal implants, etc.)
5. Do not meet the pre-screening MRI questions provided by the Center for Advanced MR Imaging (CAMRI) at BCM

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) | Every 4 hours during the tAN treatment (Days 2-6)
  The CIWA-Ar is a validated, clinician-administered scale used to assess the severity of alcohol withdrawal symptoms. The tool rates ten symptom domains-including nausea, tremor, anxiety, agitation, sweating, sensory disturbances, and orientation-to generate a total score that reflects withdrawal severity and guides clinical management. Higher scores indicate more severe withdrawal.
Average benzodiazepine use | Every 4 hours during the tAN treatment (Days 2-6)
  Benzodiazepines are commonly used to manage symptoms of alcohol withdrawal and are administered as needed based on clinical severity. Tracking benzodiazepine usage provides an indirect measure of withdrawal intensity, as higher medication requirements typically reflect more severe withdrawal symptoms, while lower usage indicates milder withdrawal.

SECONDARY OUTCOMES:
Penn Alcohol Craving Scale (PACS) | Before Day 2 and after tAN treatment on Day 6
  PACS is a validated self-report questionnaire that measures the intensity, frequency, and duration of alcohol craving over the past week. It consists of five items assessing desire to drink, anticipated likelihood of drinking, and perceived control over drinking-related thoughts. Each item is rated on a 0-6 scale, with higher total scores indicating greater craving severity.
Montgomery-Asberg Depression Scale (MADRS) | Before Day 2 and after tAN treatment on Day 6
  MADRS is a clinician-administered measure designed to assess the severity of depressive symptoms. The scale includes 10 items that evaluate core features of depression such as mood, anxiety, sleep disturbance, concentration, and suicidal ideation. Each item is scored from 0 to 6, with higher total scores indicating more severe depression.
Suicidal Behaviors Questionnaire-Revised (SBQ-R) | Before Day 2 and after tAN treatment on Day 6
  SBQ-R is a validated, self-report measure used to assess past suicidal thoughts and behaviors, as well as current risk. The questionnaire includes four items that evaluate lifetime suicidal ideation and attempts, recent ideation, threat of future suicidal behavior, and self-reported likelihood of acting on suicidal thoughts. Scores range from low to high risk, with higher scores indicating greater concern for suicidal behavior.

OTHER OUTCOMES:
Prediction of Alcohol Withdrawal Severity Scale (PAWSS) | Screening
  PAWSS is a validated clinician-administered screening tool used to identify individuals at risk for developing moderate to severe alcohol withdrawal. The scale includes 10 items assessing historical, clinical, and laboratory factors associated with withdrawal risk. A total score of 4 or higher indicates high risk for complicated withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Navid Khodaparast, PhD, Principal Investigator — Spark Biomedical, Inc.
Locations (1):
- The Menninger Clinic, Houston, Texas, United States